CLINICAL TRIAL: NCT04615078
Title: Multi-center, National, Randomized, Exploratory Study Evaluating Telemonitoring and Experimentation in Telemedicine for the Improvement of Healthcare Pathways (ETAPES Program) Compared to Standard of Care in Patients With Chronic Respiratory Failure Receiving Non-invasive Home Ventilation (e-VENT)
Brief Title: Study Evaluating Telemonitoring and Experimentation in Telemedicine for the Improvement of Healthcare Pathways (ETAPES Program) Compared to Standard of Care in Patients With Chronic Respiratory Failure Receiving Non-invasive Home Ventilation
Acronym: e-VENT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Air Liquide Santé International (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: ALMED-20-001; 2020-A02150-39 (Other: French National Agency for Medicines and Health Products Safety - ANSM (ID-RCB))
Record Dates: First submitted 2020-10-20; First posted 2020-11-04 (Actual); Last update posted 2023-06-26 (Actual); Status verified 2023-06

CONDITIONS: Chronic Respiratory Failure With Hypercapnia; Chronic Obstructive Pulmonary Disease (COPD); Obesity Hypoventilation Syndrome (OHS)
Keywords: Non-invasive ventilation; Telemonitoring; Remote Patient Management; ETAPES; Home healthcare provider; Chronic Care Connect Pneumology
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Obesity Hypoventilation Syndrome

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- "Telemonitoring" group (Experimental): Medical Telemonitoring in Non-Invasive Ventilation
  Interventions: Device: ETAPES Program
- "Standard of Care" group (No Intervention): Standard medical follow-up: standard home Non-Invasive Ventilation service, with transmission of their ventilator data without analysis leading to alerts

INTERVENTIONS:
Device: ETAPES Program — The Chronic Care Connect Pneumology is a remote medical monitoring solution, combining:
  * A technical solution for the transmission and analysis of ventilator data, leading to alerts generated by an algorithm ;
  * An organizational solution relying on a nurse call center.
  Other Names: Chronic Care Connect Pneumology Solution
  Arms: "Telemonitoring" group

SUMMARY:
The ETAPES Program, a French national Experimentation in Telemedicine for the Improvement of Healthcare Pathways, was launched in 2018 for 4 years. Its objectives were to provide a temporary public reimbursement for medical telemonitoring in order to determine the benefits for the patient and the impact on medical organization and healthcare costs. In particular, this program applies to patients suffering from hypercapnic chronic respiratory failure and requiring home non invasive ventilation (NIV). For these patients, the ETAPES program combines NIV telemonitoring and therapeutic education.

e-VENT study aims at evaluating the ETAPES program, implemented using the Chronic Care Connect™ telemonitoring solution, versus Standard of Care, on the effectiveness of home NIV, measured by average PtCO2, reflecting the level of nocturnal alveolar hypoventilation.

DETAILED DESCRIPTION:
A prospective randomized study with two arms.

The primary endpoint is the level of nocturnal alveolar hypoventilation, defined as the average PtCO2 in nocturnal capnography performed at 6th month.

Patients with hypercapnic chronic respiratory failure requiring home NIV (n=100).

Multi-center study conducted in France involving approximately 20 sites

Product under study: Chronic Care Connect Pneumology telemonitoring solution, combining:

* a technical solution for the transmission and analysis of ventilator data, with the generation of alerts by a CE-marked algorithm;
* an organizational solution relying on a nurse call center.

Study design:

* First visit: eligibility criteria confirmation; randomization to 2 groups:

  * the "Telemonitoring" group will participate in the ETAPES experimentation, with remote monitoring of their ventilator data with generation of alerts to the nurse call center, medical action if requested, and therapeutic education.
  * the "Standard of Care" group will receive standard medical follow-up, with transmission of their ventilator data without generation of alerts.
* Second visit (6th month): arterial blood gases, nocturnal capnography. Collection of medical events having occurred in the past 6 months.
* Third visit (12th month): for COPD patients only - Collection of medical events having occurred in the past 6 months.
* At the end of the study, the investigators will complete a qualitative questionnaire on their telemonitoring practice.

ELIGIBILITY:
Inclusion Criteria:

* Patient with chronic respiratory failure for whom treatment with home NIV was prescribed at inclusion or two months earlier, and whose service provider is ADEP Assistance, ADAIR Assistance, ARAIR Assistance or VitalAire,
* Patient who meets all eligibility criteria to participate in the ETAPES program, namely:

  * Patient aged 18 and over;
  * Patient receiving NIV as part of an indication recognized by the Société de Pneumologie de Langue Française and the Haute Autorité de Santé;
* Patient never before included in the ETAPES program for the remote medical monitoring of their chronic respiratory failure;
* Patient having agreed to participate in the ETAPES program with the Chronic Care Connect Pneumology solution operated by the service providers ADEP Assistance, ADAIR Assistance, ARAIR Assistance or VitalAire, in the event that they are randomized to the Remote Medical Monitoring group;
* Patient agreeing to the collection of data from their ventilator via remote transmission;
* Patient fitted with a ventilator compatible with the Chronic Care Connect Pneumology solution;
* Patient with health insurance cover;
* Patient who has signed the consent form for the study.

Exclusion Criteria:

* Patient who has any of the non-eligibility criteria for the ETAPES program:

  * Physical or mental inability to use all components of the remote medical monitoring project, as determined by the doctor wishing to include the patient in the remote medical monitoring project;
  * Patient with cancer with a life expectancy of less than 12 months estimated by the pulmonologist;
  * Patient with more than three COPD respiratory decompensations resulting in hospitalization within the previous 12 months;
  * Patient with diagnosed neuromuscular disease;
  * Estimated poor compliance or standard adherence to treatment according to the physician including the patient;
  * Patient's refusal of treatment support;
  * No permanent place of residence;
* Patient participating in another intervention research program.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2021-01-18 (Actual); Primary Completion 2022-07-25 (Actual); Study Completion 2022-07-25 (Actual)

PRIMARY OUTCOMES:
Nocturnal alveolar hypoventilation data | 6th month
  Average PtCO2, measured by transcutaneous capnography

SECONDARY OUTCOMES:
Number of medical events (consultations, hospitalizations and COPD exacerbations) related to Chronic Respiratory Failure | 6th month; 12th month
  Average number of medical events (consultations, hospitalizations and COPD exacerbations) related to Chronic Respiratory Failure per patient
Measurement of diurnal PaO2 and PaCO2 | 6th month
  Measurement of diurnal PaO2 and PaCO2 (mmHg) without NIV, in stable state at rest
S3-NIV questionnaire | Through study completion, an average estimated at around 7 months
  Questionnaire evaluating sleep, side effects and symptoms in patients on home NIV, each time the service provider visits the patient at home
DIRECT questionnaire | 1st month; 6th month
  Total health-related quality-of-life score from the DIRECT questionnaire as recommended in the ETAPES program, submitted to the patients in the month following their inclusion and in the 6th month
Quality of NIV treatment | Through study completion, an average estimated at around 7 months
  Daily data teletransmitted by ventilators throughout the follow-up period
Patient satisfaction questionnaire about Telemonitoring services | 6th month
  Questionnaire developed for the study to collect patient satisfaction about the educational component of the telemonitoring service at the end of their participation to the study

CONTACTS AND LOCATIONS:
Overall Officials: Arnaud PRIGENT, MD, Principal Investigator — Groupe Médical de Pneumologie, Polyclinique Saint Laurent - 35706 - Rennes - France
Locations (11):
- France (11):
  - Centre Hospitalier de Boulogne sur Mer, Boulogne-sur-Mer
  - Centre Hospitalier de Bligny, Briis-sous-Forges
  - Claude SCHMITZ, MD, Colmar
  - Hôpital Forcilles - Fondation Cognacq-Jay, Férolles-Attilly
  - François BUGHIN, MD - Clinique du Millénaire, Montpellier
  - Clinique FSEF Paris 16ème, Paris
  - Groupe Hospitalier Pitié Salpêtrière-Charles Foix, Paris
  - Groupe Médical de Pneumologie, Polyclinique Saint Laurent, Rennes
  - Centre Hospitalier Universitaire de Toulouse - Hôpital Larrey, Toulouse
  - Centre Hospitalier Universitaire de Tours - Hôpital Bretonneau, Tours
  - Pierre-Henri GUILLAUD, MD, Vienne

REFERENCES:
- [Derived] Prigent A, Texereau JB, Schmitz C, Ropars C, Degreef JM, Teulier M, Darne C, Lavergne F, Pasche H, Morelot-Panzini C. Real-world telemonitoring and remote support for home non-invasive ventilation to improve therapy effectiveness: the exploratory, multicentre randomised eVENT study. Thorax. 2025 Sep 15;80(10):720-729. doi: 10.1136/thorax-2024-222033. PMID 40169180